CLINICAL TRIAL: NCT00616382
Title: New Therapeutic Approaches to the Resistant Patent Ductus Arteriosus (PDA) in Low Birth Weight Neonates
Brief Title: Treating the Resistant Patent Ductus Arteriosus (PDA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Cathy Hammerman, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHPDA2
Record Dates: First submitted 2008-01-13; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-01

CONDITIONS: Patent Ductus Arteriosus
Keywords: PDA; indomethacin; pentoxifylline; Patent Ductus Arteriosus [PDA] resistant to therapy
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Indomethacin; Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepwise Indo (Experimental): Stepwise escalating doses of indomethacin, until ductal closure or maximum of 1 mg/kg/dose.
  Interventions: Drug: Indomethacin
- PTX (Experimental): Combined administration of indomethacin and pentoxifylline, an inhibitor of TNF alpha
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Indomethacin — IV indomethacin starting at a dose of 0.4 mg/kg given over 30 minutes, increased daily by increments of 0.2 mg/kg/dose and given at intervals of 12 hours until a maximum dose of 1 mg/kg is reached, or until a total indomethacin dose of 6 mg/kg has been given. Daily echocardiography will be performed to monitor the progress of ductal closure. Once echocardiographic evidence of a closed ductus is achieved, two additional doses indomethacin will be given 24 hours and 48 hours later, using the same dose used in the last indomethacin infusion.
  Arms: Stepwise Indo
Drug: Pentoxifylline — IV indomethacin will be re-started at a dose of 0.2 mg/kg to run over 30 minutes at 12 hour intervals to be given concurrently with pentoxifylline (5 mg/kg/hour to run over 6 hour once a day for a maximum of 6 days. Daily echocardiography will be performed to monitor the progress of ductal closure. Once echocardiographic evidence of a closed ductus is achieved, two additional doses indomethacin will be given 24 hours and 48 hours later and another day of pentoxifylline infusion, provided that the 6 day maximum has not yet been
  Arms: PTX

SUMMARY:
Persistent postnatal ductal patency may have significant adverse hemodynamic effects, frequently necessitating therapeutic intervention in order to facilitate ductal closure. Medical therapy for patency of the ductus arteriosus is successful mediating ductal closure in approximately 70% of treated infants. In a recent study in our population, 17% of the babies showed no ductal response to the first course of treatment and 9.4% of our study infants eventually underwent surgical ligation of the ductus after failure of medical therapeutic closure.We propose to evaluate and compare two alternate therapeutic approaches to ductal closure in babies who do not respond to initial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Inborn premature neonates admitted to the neonatal intensive care unit of the Shaare Zedek Medical Center and diagnosed as having a hemodynamically significant patent ductus arteriosus (sPDA) will be considered as potential candidates for study if/when they do not respond to initial therapy

Exclusion Criteria:

* Any baby not considered viable
* Any baby with IVH grade 3-4 of recent onset (within 3 days. [If no head ultrasound has been performed within the last 3-4 days, one should performed prior to onset of study.]
* Any baby with dysmorphic features or congenital abnormalities
* Any baby with structural heart disease other than PDA
* Any baby with documented infection,
* Any baby with thrombocytopenia (<50,000).

Ages: 2 Days to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Our primary objective in this study is to improve ductal closure rates in those infants who do not respond to a first course of therapy. | 2 years

SECONDARY OUTCOMES:
Our secondary objective is to compare the therapeutic efficacy of two very different secondary treatment protocols. | 2 years
To monitor and compare potential side effects of the two treatment approaches | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Neonatal Intensive Care Unit - Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Result] Sperandio M, Beedgen B, Feneberg R, Huppertz C, Brussau J, Poschl J, Linderkamp O. Effectiveness and side effects of an escalating, stepwise approach to indomethacin treatment for symptomatic patent ductus arteriosus in premature infants below 33 weeks of gestation. Pediatrics. 2005 Dec;116(6):1361-6. doi: 10.1542/peds.2005-0293. PMID 16322159
- [Result] Gonzalez A, Sosenko IR, Chandar J, Hummler H, Claure N, Bancalari E. Influence of infection on patent ductus arteriosus and chronic lung disease in premature infants weighing 1000 grams or less. J Pediatr. 1996 Apr;128(4):470-8. doi: 10.1016/s0022-3476(96)70356-6. PMID 8618179